CLINICAL TRIAL: NCT00776217
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Sequence, Two-Period, Single-Dose, Crossover, Bioavailability Study on Loratadine Formulations Comparing Loratadine 10 mg Orally Disintegrating Tablets of Ohm Laboratories, Inc. (A Subsidiary of Ranbaxy Pharmaceuticals Inc) With Claritin® Reditabs 10 mg Tablet (Containing Loratadine 10 mg) of Schering- Plough Healthcare Product Inc, in Healthy, Adult, Male, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study on Loratadine Orally Disintegrating Tablets 10 mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 213_LORAT_06
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence loratadine 10 mg orally disintegrating tablets fasting
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): loratadine 10 mg orally disintegrating tablets
  Interventions: Drug: loratadine 10 mg orally disintegrating tablets
- 2 (Active Comparator): loratadine 10 mg orally disintegrating tablets
  Interventions: Drug: loratadine 10 mg orally disintegrating tablets

INTERVENTIONS:
Drug: loratadine 10 mg orally disintegrating tablets

SUMMARY:
To compare the single-dose oral bioavailability of loratadine 10 mg orally disintegrating tablets of Ohm Laboratories (a subsidiary of Ranbaxy Pharmaceuticals Inc., USA) with Claritin® Reditabs® (containing loratadine 10 mg) of Schering-Plough Healthcare Product Inc., USA in healthy, adult, human male subjects under fasting condition.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomized, two-treatment, two-sequence, two-period, single-dose, crossover, bioavailability study on loratadine formulation comparing loratadine 10 mg orally disintegrating tablets of Ohm Laboratories, Inc. (a subsidiary of Ranbaxy pharmaceuticals Inc, USA) with Claritin® Reditabs® 10 mg tablet (containing loratadine 10 mg) of Schering- Plough Healthcare Product Inc, in healthy, adult, male, human subjects under fasting condition.

A single oral dose of loratadine 10 mg orally disintegrating tablets was orally administered under low light condition during each period of the study under the supervision of a trained Medical Officer. Subjects were instructed to let the tablets completely dissolve on the tongue before swallowing the saliva and then, 240 mL of water was administered 30 seconds after drug administration.

During the course of the study safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical parameters and urine analysis) at baseline. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

A total of 80 subjects were randomized to receive a single oral dose of the test or reference formulation for loratadine 10 mg. Seventy-four subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years.
* Were neither overweight nor underweight for the corresponding height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* Had history of allergy to loratadine.
* Had history of hypertension.
* Had any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Had history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes or glaucoma.
* Had presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Had presence of values which were significantly different from normal reference ranges and/or judged clinically significant for hemoglobin, total white blood cells count, differential WBC count or platelet count.
* Was positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Had presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Had clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
* Had clinically abnormal ECG or Chest X-ray.
* Had history of any psychiatric illness, which might impair the ability to provide written informed consent
* Was a regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* Had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Used any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Had participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html